#### Janssen Pharmaceutical K.K. \*

## Statistical Analysis Plan for Primary Analysis, and Final Analysis

A Phase 2a, Multicenter, Open-label Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Combination Treatment of AL-335, Odalasvir, and Simeprevir in Japanese Subjects With Chronic Hepatitis C Genotype 1 or 2 Virus Infection, With or Without Compensated Cirrhosis who are Direct-acting Antiviral Treatment-naïve

## Protocol 64294178HPC2003; Phase 2a

AL-335, Odalasvir, TMC435(simeprevir)

\*This study is being conducted by Janssen Pharmaceutical K.K. in Japan. The term "sponsor" is used throughout the protocol to represent Janssen Pharmaceutical K.K.

Status: Approved

Date: 8 June 2018

**Prepared by:** Janssen Pharmaceutical K.K. **Document No.:** EDMS-ERI-164033457

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

## **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | 2 |
|---|---|---|
| ABBRI | EVIATIONS | 4 |
| | NTRODUCTION | |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | |
| 1.2.1. | Endpoints | |
| 1.2.1. | Statistical Hypotheses for Trial Objectives | |
| 1.3.<br>1.4. | | |
| 1. <del>4</del> .<br>1.5. | Sample Size Justification | |
| | • | |
| | SENERAL ANALYSIS DEFINITIONS | |
| 2.1. | Visit Windows and Phase Definition | |
| 2.2. | Pooling Algorithm for Analysis Centers | |
| 2.3. | Analysis Sets | |
| 2.4. | Definition of Subgroups | 10 |
| | SUBJECT INFORMATION | |
| 3.1. | Demographics and Baseline Characteristics | |
| 3.2. | Disposition Information | 11 |
| 3.3. | Treatment Adherence | 12 |
| 3.4. | Extent of Exposure | 12 |
| 3.5. | Protocol Deviations | |
| 3.6. | Prior and Concomitant Medications | 12 |
| 3.7. | Medical History | 13 |
| 4. E | FFICACY | 13 |
| 4.1. | Level of Significance | 13 |
| 4.2. | Data Handling Rules | 13 |
| 4.3. | Efficacy Endpoints | 13 |
| 4.3.1. | Definitions | 14 |
| 4.3.2. | Analysis Methods | 17 |
| 4.3.3. | Treatment Stopping Rules | 18 |
| 5. V | /IROLOGY | 19 |
| 5.1. | Virology Assessments | 19 |
| 5.1.1. | Viral strain typing | |
| 5.1.2. | Viral sequencing | |
| 5.2. | Virology Definitions | |
| 5.3. | Virology Time Points and Samples | 20 |
| 5.4. | Virology Analyses | |
| 5.4.1. | HCV geno/subtype analyses | |
| 5.4.2. | Resistance analyses | 2 |
| 5.4.2.1 | | |
| 5.4.2.2 | | |
| 5.4.2.3 | . Over the Study Period | 2 |
| 6. S | SAFETY | 2' |
| 6.1. | Adverse Events | |
| 6.1.1. | Definitions | |
| 6.1.2. | Analysis Methods | |
| 6.2. | Clinical Laboratory Tests. | |
| 6.2.1. | Definitions | |
| 6.2.2. | Analysis Methods | |
| 6.3. | Vital Signs and Physical Examination Findings | |
| | G | |

## Statistical Analysis Plan 64294178HPC2003

| 6.3.1. | Definitions | 25 |
|---|---|---|
| 6.3.2. | Analysis Methods | |
| 6.4. | Electrocardiogram | |
| 6.4.1. | Definitions | |
| 6.4.2. | Analysis Methods | <mark>27</mark> |
| 6.5. | Echocardiography | |
| 6.5.1. | Definitions | <mark>2</mark> 8 |
| 6.5.2. | Analysis Methods | <mark>2</mark> 8 |
| 6.6. | Patient Profiles | <mark>2</mark> 9 |
| 7. F | PHARMACOKINETICS/PHARMACODYNAMICS | 20 |
| 7. г<br>7.1. | PharmacokineticsPharmacobinamics | |
| 7.1.<br>7.2. | Immune Response | |
| 7.2.<br>7.3. | Pharmacodynamics | |
| 7.4. | Pharmacokinetic/Pharmacodynamic Relationships | |
| ATTA | CHMENTS | 30 |
| ΔΡΡΕΙ | NDIX 1: PHASE ALLOCATION/COMBINING AES | 3( |
| AII L | TOTAL RECOGNICION/COMBINING ACCUMENTATION AC | |
| APPE | NDIX 2A: SEARCH TERMS FOR EVENTS OF SPECIAL/CLINICAL INTEREST | 32 |
| APPE | NDIX 2B: RASH - SMQ19.1 | 33 |
| APPE | NDIX 3: CARDIAC EVENTS - SMQ19.1 | 34 |

#### **ABBREVIATIONS**

ADaM Analysis Data Model Adverse Event ΑE **Body Mass Index** BMI Change from Baseline **CFB** Clinical Trial Protocol CTP DAA **Direct-Acting Antivirals** DRC Data Review Committee **ECG** Electrocardiogram

ECHO Echocardiogram / Echocardiography

eCRF Electronic Case Report Form

EOT End Of Treatment
HCV Hepatitis C Virus
IA Interim Analysis
ITT Intent-To-Treat
LV Left Ventricular

LVEF Left Ventricular Ejection Fraction

NAP Not Applicable ODV Odalasvir PT Preferred Term

QD Quaque Die, Once Daily RNA Ribonucleic Acid SAE Serious Adverse Event SAP Statistical Analysis Plan SI Standard International

SMV Simeprevir

SOC System Organ Class WHO World Health Organization

#### 1. INTRODUCTION

This 64294178HPC2003 Statistical Analysis Plan (SAP) covers Cut-Off Analysis, Primary Analysis and Final Analysis. It contains definitions of analysis sets, derived variables and statistical methods for the analysis. Separate document for DPS is also provided. A separate SAP was written for the Data Review Committee (DRC) analyses.

Please refer to the study protocol for the background for the study.

## 1.1. Trial Objectives

## **Primary Objectives**

• To evaluate the safety and tolerability of a combination treatment of AL-335, ODV, and SMV for 8 weeks in DAA-naïve Japanese subjects with genotype 1 or 2 chronic HCV infection without cirrhosis and for 12 weeks in DAA-naïve Japanese subjects with genotype 1 or 2 chronic HCV infection with compensated cirrhosis.

### **Secondary Objectives**

- To evaluate the PK of AL-335 (and metabolites), ODV, and SMV in plasma in Japanese subjects with genotype 1 or 2 chronic HCV infection with or without compensated cirrhosis who are DAA-naïve.
- To evaluate the efficacy, ie, SVR4, SVR12, and SVR24, of a combination treatment with AL-335, ODV, and SMV for 8 weeks in DAA-naïve Japanese subjects with genotype 1 or 2 chronic HCV infection without cirrhosis and for 12 weeks in DAA-naïve Japanese subjects with genotype 1 or 2 chronic HCV infection with compensated cirrhosis.
- To evaluate on-treatment viral kinetics in an 8 or 12-week treatment regimen containing AL-335, ODV, and SMV in subjects who are DAA- naïve.
- To evaluate the incidence of on-treatment failure during an 8 or 12-week treatment regimen containing AL-335, ODV, and SMV in subjects who are DAA-naïve.
- To evaluate the incidence of viral relapse after an 8 or 12-week treatment regimen containing AL-335, ODV, and SMV in subjects who are DAA-naïve.

## **Exploratory Objectives**

- To explore relationships of exposure of AL-335 (and metabolites), ODV, and SMV with SVR and safety.
- To evaluate the impact of the patient and disease characteristics at baseline on SVR, including but not limited to prior treatment history, IL28B genotype, presence of cirrhosis, HCV RNA level, and HCV geno/subtype.
- To evaluate the impact of the presence of HCV NS3/4A, NS5A, and/or NS5B polymorphisms at baseline on treatment outcome.
- To assess the emergence of resistant variants in subjects not achieving SVR.

## 1.2. Trial Design

This is a Phase 2a, multicenter, open-label study. It consists of a 6-week Screening Period, followed by the 8-week or 12-week Treatment Period, and the 24-week Posttreatment Follow-up Period.

Approximately 20 DAA-naïve chronic HCV genotype 1 or 2-infected subjects without cirrhosis will be assigned to Cohort 1, and approximately 20 DAA-naïve chronic HCV genotype 1 or 2-infected subjects with compensated cirrhosis will be assigned to Cohort 2.

- Cohort 1 (N=20, chronic hepatitis C without cirrhosis):
   AL-335 800 mg once daily + ODV 25 mg once daily + SMV 75 mg once daily for 8 weeks
- Cohort 2 (N=20, chronic hepatitis C with compensated cirrhosis):

AL-335 800 mg once daily + ODV 25 mg once daily + SMV 75 mg once daily for 12 weeks

To conduct this study carefully in light of securing subjects' safety, after 6 subjects in Cohort 1 completed the Week 4 visit, DRC will review all available relevant safety data to make a decision about start of dosing in Cohort 2.

Further trial design details are available in the protocol.

### 1.2.1. Endpoints

### **Primary Endpoint**

Safety data, including but not limited to adverse events (AEs), 12-lead electrocardiograms (ECGs), echocardiograms, and clinical laboratory results (including chemistry, hematology, and urine).

## **Secondary Endpoints**

- PK parameters for AL-335 (and metabolites), ODV, and SMV in plasma
- The proportion of subjects who have an SVR4, SVR12, and SVR24
- The proportion of subjects with viral relapse
- The proportion of subjects with on-treatment failure
- The proportion of subjects with on-treatment virologic response:
  - HCV RNA not detected
  - HCV RNA <LLOQ</li>
- Time to achieve HCV RNA not detected or HCV RNA <LLOQ</li>

### **Exploratory Endpoints**

• The effect of the presence or absence at baseline of HCV NS5A, NS5B, and/or NS3/4A polymorphisms on treatment outcome

- The changes in the HCV NS3/4A, NS5A and/or NS5B sequences in subjects not achieving SVR
- Impact of baseline condition on SVR (including but not limited to prior treatment history, IL28B genotype, presence of cirrhosis, HCV RNA level, and HCV geno/subtype)

## 1.3. Statistical Hypotheses for Trial Objectives

The study is hypothesis-generating. No formal hypothesis will be tested

## 1.4. Sample Size Justification

Since this is an exploratory study, no formal sample size calculation has been performed.

With a total sample size of 40 subjects, the probability to observe an AE with an incidence of 10.0% is 99.0%. The probability to observe an AE with an incidence of 1.0%, 2.5%, and 5.0% is 33.0%, 64.0%, and 87.0%, respectively. With 20 subjects per cohort, the probability to observe an AE with an incidence of 10.0% is 88.0%. The probability to observe an AE with an incidence of 1.0%, 2.5%, and 5.0% is 18.0%, 40.0%, and 64.0%, respectively in a cohort.

With an expected SVR rate of 90.0%, and 40 subjects in 2 cohorts combined, the corresponding 95%, 2-sided confidence interval (CI) is 76.3% to 97.2%. With 95.0% SVR, the corresponding 95% CI ranges from 83.1% to 99.4%. With an expected SVR rate of 90.0%, and 20 subjects per cohort, the corresponding 95%, 2-sided CI is 68.3% to 98.8%. With 95.0% SVR, the corresponding 95% CI ranges from 75.1% to 99.9% in a cohort.

Therefore, a total sample size of approximately 40 subjects is considered sufficient to explore the safety and efficacy of the combination regimen consisting of AL-335, ODV, and SMV in this study from a clinical point of view.

## 1.5. Randomization and Blinding

Randomization and Blinding will not be used as this is an open-label study. Subjects will be assigned to a treatment cohort based on the presence or absence of cirrhosis.

### 2. GENERAL ANALYSIS DEFINITIONS

#### 2.1. Visit Windows and Phase Definition

Phases will be constructed as indicated in Table 1 and Table 2.

**Table 1: Phase Definition Part 1** 

| Cohort | W-6 | D1 | D2 | D3 | W1 | W2 | W3 | W4 | W6 | W8 | - | - | W4<br>FU | W8<br>FU | W12<br>FU | W18<br>FU | W24<br>FU |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 | Scr. | | | AL-33 | 35 + O | DV + S | SMV 8 | weeks | | | - | - | | Fo | ollow up | ) | |
| Weeks | W-6 | D1 | D2 | D3 | W1 | W2 | W3 | W4 | W6 | W8 | W10 | W12 | W4<br>FU | W8<br>FU | W12<br>FU | W18<br>FU | W24<br>FU |
| Cohort 2 | Scr. | | | | AL-3 | 35 + O | DV + | SMV 1 | 2 wee | ks | | | | Fo | ollow up | ) | |

| Table 2: | Phase Definition Part 2 | |
|---|---|---|
| Trial phase | Start date | End date |
| Screening | Minimum of Date of signing the informed | 1 day before first study drug administration |
| (phase 0) | consent and Date of the first screening visit | |
| Treatment | Date of first study drug administration | Date of last study drug intake + 3 days |
| (phase 1) | | |
| Follow-up | Phase 1 end date +1 day | Trial termination date (date of last contact) |
| (phase 2) | | |

<u>Date of First Study Drug Administration</u>: In the above computations, missing data for first study drug intake may be imputed as the date of baseline visit.

<u>Date of Last Study Drug Administration:</u> In the above computations, missing data for last study drug intake may be imputed for cut-off analysis and subjects discontinued as follows:

- 1. Cut-off analyses: Date of Last Study Drug Intake = Min (Data cutoff date, Date of baseline visit + 8 or 12 weeks depending on cohort).
- 2. Date of Last Study Drug Intake =
  - a. Date of the early treatment withdrawal visit, if nonmissing otherwise
  - b. Date of 1<sup>st</sup> available Follow-up visit 28, if nonmissing otherwise
  - c. Date of last contact.

#### Reference date is defined as:

- Screening and Treatment Phases: Reference date = Date of first study drug intake (if nonmissing), otherwise date of baseline visit.
- Follow-up Phase: Reference date = Start Date of follow-up phase.

The number of days in the phase (Relative day) is defined as:

- Visits on or after the reference date: Relative day = visit date reference date+1
- Visits before the reference date: Relative day = visit date reference date
- Actual EOT visit is defined as the last visit in the Treatment phase.

All visits (regardless of the investigated parameter) will be allocated to analysis time points based on the number of days in phase (relative day) as indicated in Table 3.

**Table 3: Visit Windows** 

| Trial phase | Target day | Analysis time point (numeric version) | Analysis time point | Time interval (Relative day) |
|---|---|---|---|---|
| Cohort 1 | | | | |
| Screening phase | + ∞ | -1 | Screening | <0 |
| Treatment | 1 | 0 | Baseline <sup>a</sup> | <=1 |
| phase | 2 | 0.2 | Day 2 | [2,2] |
| | 3 | 0.3 | Day 3 | [3,5] |
| | 7 | 1 | Week 1 | [6,11] |
| | 14 | 2 | Week 2 | [12,18] |
| | 21 | 3 | Week 3 | [19,25] |
| | 28 | 4 | Week 4 | [26,35]<br>[36,49] |
| | 42<br>56 | 6<br>8 | Week 6<br>Week 8 | $[50, +\infty]$ |
| | last visit while on<br>study therapy or within<br>3 days after the day of<br>last dose | 999 | EOT | [50, + \omega] |
| Follow-up phase | 25 | 16 | Follow-Up Week 4 | [1,39] |
| phase | 53 | 20 | Follow-Up Week 8 | [40,67] |
| | 81 | 24 | Follow-Up Week 12 | [68,102] |
| | 123 | 30 | Follow-Up Week 18 | [103,144] |
| | 165 | 36 | Follow-Up Week 24 | [145, +∞] |
| Cohort 2 | | | | |
| Screening phase | -∞ | -1 | Screening | <0 |
| Treatment | 1 | 0 | Baseline <sup>a</sup> | <=1 |
| phase | 2 | 0.2 | Day 2 | [2,2] |
| | 3 | 0.3 | Day 3 | [3,5] |
| | 7 | 1 | Week 1 | [6,11] |
| | 14 | 2 | Week 2 | [12,18] |
| | 21 | 3 | Week 3 | [19,25] |
| | 28 | 4 | Week 4 | [26,35] |
| | 42<br>56 | 6 | Week 6 | [36,49] |
| | 70 | 8<br>10 | Week 8<br>Week 10 | [50,63]<br>[64,77] |
| | 84 | 12 | Week 12 | $[78, +\infty]$ |
| | last visit while on<br>study therapy or within<br>3 days after the day of<br>last dose | 999 | EOT | [70, 1 ∞] |
| Follow-up<br>phase | 25 | 16 | Follow-Up Week 4 | [1,39] |
| phase | 53 | 20 | Follow-Up Week 8 | [40,67] |
| | 81 | 24 | Follow-Up Week 12 | [68,102] |
| | 123 | 30 | Follow-Up Week 18 | [103,144] |
| | 165 | 36 | Follow-Up Week 24 | $[145, +\infty]$ |

### Note:

Target day in follow up phase equals target day in the protocol minus 3 days due to definition of start of follow-up phase.

If two visits fall within the same interval, the last measurement within the interval will be used for descriptive statistics/tabulations per time point and graphics in order to have only one evaluation per subject per analysis time point. If two measurements occur on the same day, the measurement with highest sequence number will be used. Listings will include all values.

## 2.2. Pooling Algorithm for Analysis Centers

No pooling of analysis subcenters will be performed in this study.

## 2.3. Analysis Sets

Safety Analysis Set: All enrolled subjects who received at least 1 dose of study drug (AL-335, ODV, or SMV).

Full Analysis Set (FAS): All enrolled subjects who received at least 1 dose of study drug (AL-335, ODV, or SMV) and have at least 1 postbaseline efficacy measurement.

*Non-VF Excluded Set*: All FAS subjects excluding subjects with early treatment discontinuation due to nonvirologic reasons or missing data at SVR4, SVR12, or SVR24 time points.

All analyses except for efficacy, and virology analyses will be done on safety analysis set. The efficacy analyses will be performed on full analysis set. Selected virology analyses will be using non-VF excluded set as needed. Demographic and baseline characteristics should be done on the safety.

## 2.4. Definition of Subgroups

The subgroups will be used to perform analyses on efficacy endpoints are:

- Age category  $[\le 65; > 65]$
- BMI [<25; ≥25]
- IL28B genotype (CC, CT, TT); and also (CC, non-CC)
- Gender (male, female)
- HCV geno/subtype (1a, 1b, 1other, 1a with Q80K, 1a without Q80K, 2a, 2b, 2c, 2other)
- baseline HCV RNA categories (<6,000,000 IU/mL, ≥6,000,000 IU/mL)

The subgroups will be used to perform analyses on safety endpoints are:

- Age category [≤65; >65]
- BMI [<25; ≥25]
- Gender (male, female)

#### 3. SUBJECT INFORMATION

### 3.1. Demographics and Baseline Characteristics

Descriptive statistics or tabulation will be provided, in addition to listings, for the following parameters:

## **Demographic parameters**

• Gender (male, female)

- Age at screening (years)
- Age at screening (years, categories:  $\leq 45$ ;  $\geq 45 \leq 65$ ;  $\geq 65$ )
- Race (Asian)
- Ethnicity (Not Hispanic or Not Latino)
- Weight at baseline (kg)
- BMI at baseline = weight (at baseline, in kg)/ (height (at screening, in meters))<sup>2</sup>, rounded to 1 decimal (although available in the raw data, BMI will be recalculated from weight and height)
- BMI at baseline (categories:  $\langle 25, 25 \langle 30, \geq 30 \rangle$ )

### **Baseline disease characteristics**

- baseline HCV RNA (original and log<sub>10</sub> units)
- baseline HCV RNA categories (<6,000,000 IU/mL, ≥6,000,000 IU/mL)
- HCV geno/subtype 1a, 1b, 1other, 1a with Q80K, 1a without Q80K, 2a, 2b, 2c, 2other
- Prior IFN with or without RBV taken (Yes or No)
- IL28B subtype (CC, CT, TT)
- For subjects with Fibroscan Results:
  - Fibroscan Metavir Fibrosis Result (kPa)
  - Fibroscan Metavir Fibrosis stage (F0/F1, F2, F3, F4)
- For subjects with Biopsy Results (Each subject has either Metavir or Ishak scoring):
  - Biopsy Metavir Fibrosis stage (F0/F1, F2, F3, F4)
  - Metavir Inflammation grade (A0, A1, A2, A3)
  - Biopsy Ishak Fibrosis stage (0, 1, 2, 3, 4, 5, 6)
  - Ishak Inflammation grade (1-3, 4-8, 9-12, 13-18)
- Time since diagnosis (years) (= (baseline date date of diagnosis + 1)/365.25, rounded to 1 decimal)

### 3.2. Disposition Information

Tabulations will be provided for the following disposition information:

- Number of subjects screened, enrolled and treated
- Number of subjects with a visit per analysis time point
- Number of subjects prematurely discontinuing any single study medication and the reason for discontinuation (obtained from the treatment disposition page of the electronic case report form [eCRF])

• Number of subjects prematurely discontinuing the trial and the reason for discontinuation. Reasons for discontinuation are obtained from the trial disposition page of the eCRF.

### 3.3. Treatment Adherence

For each of the three drugs (AL-335, Odalasvir, SMV), the actual amount (actual dose over actual treatment duration) of study drug relative to the planned cumulative total dose (planned dose over planned duration) will be summarized.

For each drug, the number (%) of subjects with  $\leq 3$  and > 3 consecutive days of dose interruption will be tabulated. The number of subjects without a dose interruption will also be tabulated. Summary statistics for the total number of days of dose interruption for subjects with at least one day of dose interruption will also be tabulated. Further, for each drug, the number (%) of subjects with  $\leq 3$ ,  $4 - \leq 6$ , and  $\geq 6$  cumulative days of dose interruption will be tabulated.

## 3.4. Extent of Exposure

Treatment duration (in weeks) is derived as follows for each of the three drugs (AL-335, Odalasvir, SMV):

• (Last date of exposure – first date of exposure + 1) / 7

Note: treatment interruptions will not be taken into account for the above definition.

Treatment duration and total dose received will be summarized descriptively by treatment cohort. Treatment duration for subjects who did not complete treatment will also be summarized descriptively by treatment cohort.

#### 3.5. Protocol Deviations

All major protocol deviations will be tabulated. Additionally, all protocol deviations (major and minor) will be listed. Major protocol deviations that may affect the assessment of efficacy will be flagged in the listing.

#### 3.6. Prior and Concomitant Medications

Prior medications will be tabulated by treatment cohort. Concomitant medications will be tabulated by treatment cohort and by phase. Concomitant medications are allocated to phases based on their start and stop date. The concomitant medications will be allocated to a phase during which they were applied. A concomitant medication can be allocated to more than one phase.

Incomplete dates (ie, day and/or month and/or year missing):

• In case of a partial start date, the therapies are allocated to the phases using the available partial information, no imputation is done. If, for instance, for a therapy start date only month and year is available, these data are compared with the month and year info of the phases.

- In case of a completely missing start date, the therapy is considered as having started before the trial
- In case of a completely missing end date, the therapy is considered as ongoing at the end of the trial

## 3.7. Medical History

Frequency tabulations of medical history will be provided. A listing of medical history will also be provided.

#### 4. EFFICACY

## 4.1. Level of Significance

No significance testing will be performed in this study. However, a 95% CI will be constructed around the proportion of subjects with SVR and other virologic response parameters.

## 4.2. Data Handling Rules

Plasma HCV RNA will be determined using an in vitro nucleic acid amplification test for the quantification of HCV RNA in human plasma using a sensitive assay (COBAS® AmpliPrep/COBAS® TaqMan® HCV Test v2.0, lower limit of quantification [LLOQ] = limit of detection [LOD] = 15 IU/mL). HCV RNA determination will be performed at a central laboratory.

Before performing continuous analyses or log transformations, HCV RNA results of '<LLOQ IU/mL HCV RNA DETECTED' will be converted to LLOQ-1 IU/mL and 'HCV RNA NOT DETECTED' will be converted to LOD-2 IU/mL.

Note: We subtract 2 from the LOD to distinguish between '<LLOQ IU/mL HCV RNA DETECTED' and '<HCV RNA NOT DETECTED' in all cases, as the LLOQ could equal the LOD.

For the purpose of sensitivity analysis, missing HCV RNA data for subjects who discontinued early will be imputed using Last Observation Carry Forward(LOCF).

## 4.3. Efficacy Endpoints

The efficacy endpoints are listed as below:

- The proportion of subjects who have an SVR4, SVR8, SVR12, SVR18 and SVR24;
- The proportion of subjects with viral relapse
- The proportion of subjects with on-treatment failure
- The proportion of subjects with on-treatment virologic response (HCV RNA Not Detected or HCV RNA <LLOQ)
- Time to achieve on-treatment virologic response (HCV RNA Not Detected or HCV RNA <LLOQ)

#### 4.3.1. Definitions

#### **SVRx** is defined as follows:

- 1=success:
  - at the time point of SVR
    - HCV RNA Not Detected or
    - o HCV RNA <LLOQ and
      - ♦ the sample is a confirmation\* sample or
      - the sample is the last available HCV RNA measurement or
      - ♦ at the next available measurement, HCV RNA Not Detected or HCV RNA <LLOQ Detected</p>
    - $\circ \ge LLOQ$  quantifiable and
      - the sample is not a confirmatory sample\* and
      - not the last available measurement in the study and
      - ◆ a next measurement is available and HCV RNA Not Detected or HCV RNA
         <LLOQ for this next measurement</li>
- 0= failure: otherwise
- \* Confirmed means that the criterion should be fulfilled at 2 or more consecutive time points or at the last observed time point.

Add 'The LLOQ for the HCV RNA COBAS® AmpliPrep/COBAS® TaqMan® Test v2.0, used in this study, is 15 IU/mL.' as a footnote.

### Time point of SVR24 is defined as:

- 24 weeks after the actual EOT (Select the measurement in the SVR24 analysis window. If >1 measurements are present in this window then select the one latest in time.)
- or, if not available, the first available measurement at least 24 weeks after the actual EOT (ie, the first available measurement after the SVR24 analysis window)
- or, if not available, the last measurement available in the SVR18 analysis window, on condition that the time point of SVR24 has been reached
- or, if not available, the last measurement available in the SVR12 analysis window, on condition that the time point of SVR24 has been reached
- or, if not available, the subject is considered to have not achieved SVR24.

### Time point of SVR18 is defined as:

• 18 weeks after the actual EOT (Select the measurement in the SVR18 analysis window. If >1 measurements are present in this window then select the one latest in time.)

- or, if not available, the first available measurement at least 18 weeks after the actual EOT (ie, the first available measurement after the SVR18 analysis window)
- or, if not available, the last measurement available in the SVR12 analysis window, on condition that the time point of SVR18 has been reached
- or, if not available, the subject is considered to have not achieved SVR18.

## **Time point of SVR12** is defined as:

- 12 weeks after the actual EOT (Select the measurement in the SVR12 analysis window. If >1 measurements are present in this window then select the one latest in time.)
- or, if not available, the first available measurement at least 12 weeks after the actual EOT (ie, the first available measurement after the SVR12 analysis window)
- or, if not available (ie, no measurement at least 12 weeks after the actual EOT), the subject is considered a failure.

Time point SVR4 and time point SVR8 are defined similarly as time point SVR12 as above.

### **Evaluated in the treatment phase:**

On-Treatment Virologic Response is defined as follows:

- 0 = HCV RNA result not satisfying a specified threshold
- 1 = HCV RNA result satisfying a specified threshold

The following thresholds will be considered at any time point during treatment:

- HCV RNA Not Detected
- HCV RNA < lower limit of quantification (LLOQ) (detected or not detected)

Note: virologic response will always be calculated as on-treatment response; therefore, the denominator will only include those subjects with valid on-treatment HCV RNA per analysis time point.

Other definitions of virologic response:

vRVR (Very Rapid Virologic Response): HCV RNA Not Detected at Week 2 of treatment (the denominator for the proportion of subjects with vRVR will be the number of subjects who have a nonmissing Week 2 measurement while on therapy (or within 3 days of the date of last dose))

RVR (Rapid Virologic Response): HCV RNA Not Detected at Week 4 of treatment (the denominator for the proportion of subjects with RVR will be the number of subjects who have a nonmissing Week 4 measurement while on therapy (or within 3 days of the date of last dose))

Time to On-treatment Virologic Response is defined as: The number of days since the first day of medication intake until the first day that the threshold (HCV RNA Not Detected or HCV RNA <LLOQ) was achieved.

**On-treatment Failure** is defined as: Subjects who do not achieve SVR12, with confirmed HCV RNA  $\geq$ LLOQ at the actual EOT. Includes subjects with:

- **viral breakthrough**, defined as a confirmed\* increase of >1.0 log<sub>10</sub> IU/mL in HCV RNA from nadir, or confirmed HCV RNA >2.0 log<sub>10</sub> IU/mL in subjects whose HCV RNA had previously been <LLOQ while on treatment.
- other with confirmed HCV RNA ≥LLOQ at the actual EOT (eg, completed study drug treatment, discontinued due to AEs, withdrawal of consent).

\*Confirmed means that the criterion should be fulfilled at 2 or more consecutive time points or at the last observed time point.

The proportion of subjects with a viral breakthrough is defined as follows:

- 0 = subject has not had a viral breakthrough (see definition above) up to the considered time point
- 1 = subject has a viral breakthrough at the considered timepoint or has had a viral breakthrough before (regardless of the HCV RNA result at the considered time point)

### **Evaluated in the treatment and follow-up phases:**

*Failure:* subjects not achieving SVR12 including:

- In the treatment phase: On-treatment failure (see above)
- In the follow-up phase: Posttreatment failure, includes subjects with:
  - Viral relapse after completed treatment
  - Viral relapse after premature discontinuation of treatment
  - Missing HCV RNA at timepoint of SVR12.

<u>Type of failure</u>: if more than 1 type of failure occurs, the order as presented below should be respected:

- 1. Viral Relapse
- 2. Viral breakthrough
- 3. Confirmed HCV RNA ≥LLOQ at EOT
- 4. Missing at timepoint of SVR12

## **Evaluated in the follow-up phase:**

### **Viral relapse** is defined as follows:

## 1 = viral relapse

Subject is not achieving SVR12 (see above)

and

o Subject is not an on-treatment failure (see above)

and

- o Post treatment HCV RNA measurement fulfill one of the following conditions:
- o at least 2 consecutive measurements are ≥ LLOQ IU/mL quantifiable

or

- o the last available measurement is  $\geq$  LLOQ IU/mL quantifiable
- 0 = no viral relapse: at least one posttreatment measurement available and not a viral relapse
- 2 = no posttreatment HCV RNA measurements available

Note: viral relapse will only be assessed for those subjects with no on-treatment failure. The denominator will only include those subjects with values 0 and 1.

### Late Viral relapse is defined as follows:

#### 1 = late viral relapse

Subject is achieving SVR12 (see above)

and

- Post treatment HCV RNA measurement beyond the SVR12 time point fulfill one the following conditions:
  - ♦ at least 2 consecutive measurements are ≥ LLOQ IU/mL quantifiable

or

- o the last available measurement is  $\geq$  LLOQ IU/mL quantifiable
- 0 = no late viral relapse: at least one measurement after the time point of SVR12 available and not a late viral relapse.
- 2 = no measurement after time point of SVR12 available.

Note: late viral relapse will only be assessed for those subjects with no on-treatment failure and no viral relapse. The denominator will only include those subjects with values 0 and 1.

### 4.3.2. Analysis Methods

All efficacy analyses will be using the full analysis set by cohort.

Descriptive statistics (n, mean (SD), median, interquartile ranges and ranges) per time point by treatment cohort for the continuous parameters (actual values and change from baseline in log<sub>10</sub> for HCV RNA). Corresponding listings will be presented. Mean (SD) plots will be produced for actual values and change from baseline in log<sub>10</sub> for HCV RNA by treatment cohort.

Tabulations (numbers, proportions and 95% CI) per cohort and time point for SVR4, SVR8, SVR12, SVR18 and SVR24 will be provided. The sensitivity analysis with LOCF applied to missing HCV RNA data will also be performed. The number and proportion of subjects with ontreatment failure and on-treatment virologic response will be tabulated by cohort and overall. Corresponding listings will be presented.

For time to on-treatment virologic response, descriptive statistics (n, mean (SD), median, interquartile ranges and ranges) by treatment cohort will be tabulated.

Subgroup analyses as defined in Section 2.4 will be performed for the selected endpoints.

In addition, the reason for failure will be explored by type of failure (see definition of failure above). If more than one type of failure occurs, the order as presented below should be respected:

- 1. viral relapse
- 2. viral breakthrough
- 3. confirmed HCV RNA ≥LLOQ at the actual EOT
- 4. missing at time point of SVR12

## 4.3.3. Treatment Stopping Rules

All study drugs will be discontinued for any subject with viral breakthrough (see the definition in Section 4.3.1). Additionally, an individual subject may stop one or all study drugs if a specific toxicity is met (see Section 6.4 of the protocol for full details).

The occurrence of any one of the following treatment-emergent events in any ongoing study using ODV at therapeutic doses:

- 2<sup>nd</sup> degree Mobitz Type 2 or 3<sup>rd</sup> degree heart block;
- drop in EF by  $\ge 10$  points with absolute EF < 50%;
- a cardiac event that is serious, severe or life-threatening;

will lead to stop of recruitment and dosing in all subjects in the current study if adjudicated by the DRC to be at least possibly related to the study regimen. Such event(s) will be reported to the sponsor medical monitor within 24 hours. Upon this notification, a safety assessment of the event by the DRC will take place within 48 hours and the outcome of the assessment and its associated action towards the study will be reported to Health Authorities and Ethics Committees in compliance with safety reporting regulations, as applicable.

### 5. VIROLOGY

## 5.1. Virology Assessments

## 5.1.1. Viral strain typing

The HCV geno/subtype is determined at screening for study eligibility/stratification using the HCV LiPA v2.0 test and in case no result is obtained the NS5B-based test is used as reflex. In addition, the HCV geno/subtype is determined at baseline for efficacy and virology analyses using the NS5B-based test. In case no result at baseline is obtained, the screening results are used for efficacy and virology analyses.

## 5.1.2. Viral sequencing

The HCV NS3/4A, NS5A and NS5B regions are sequenced using Next Generation Sequencing (1% read frequency cut-off) in all subjects at baseline and postbaseline in subjects not achieving SVR, focusing on the time of virologic failure and the end of study.

## 5.2. Virology Definitions

**Baseline polymorphisms** are defined as amino acid differences from a HCV reference strain with a read frequency  $\geq 15\%$ . The reference strains used for the genotypes included in the study are shown in Table 4.

**Table 4:** Reference Strain for Genotypes

| Genotype | Reference Strain<br>(GenBank Accession ID) |
|---|---|
| 1a | H77 (NC_004102) |
| 1b | Con1 (AJ238799) |
| Other genotype 1 subtypes or subtype unknown | H77 (NC_004102) |
| 2 | JFH-1 (AB047639) |

**Treatment-emergent substitutions** are defined as amino acids detected postbaseline  $\geq 15\%$  and not detected (ie, <1%) at baseline.

**Treatment-enriched substitutions** are amino acids detected at baseline with a read frequency  $\geq 1\%$  and  $\leq 15\%$ , and with an increase in read frequency of at least 15% postbaseline.

**Return to Baseline** is defined as a treatment-emergent substitution which is no longer detected (ie <1%) at end of study, but instead the baseline amino acid is observed.

**Resistance-associated substitutions (RASs)** are amino acids present at baseline or postbaseline at the positions of interest (see below) in the sequenced regions which are known to confer resistance to one of the drugs. Of note, not all amino acids at the positions of interest are RASs.

## **HCV NS3 positions of interest:**

- List of 18 positions associated with resistance to NS3/4A protease inhibitors: 36, 41, 43, 54, 55, 80, 107, 122, 132, 138, 155, 156, 158, 168, 169, 170, 174 and 175
- List of 8 positions associated with resistance to SMV: 43, 80, 122, 132, 155, 156, 168 and 170

### **HCV NS5A positions of interest:**

- List of 18 positions associated with resistance to NS5A inhibitors: 6, 21, 23, 24, 28, 29, 30, 31, 32, 37, 38, 52, 54, 58, 62, 64, 92, and 93
- List of 8 position associated with resistance to ODV: 28, 29, 30, 31, 32, 58, 92, and 93

#### **HCV NS5B positions of interest:**

• List of 9 positions associated with resistance to nucleotide analog NS5B polymerase inhibitors: 96, 142, 159, 223, 226, 282, 316, 320, and 321

**Virologic Failure (VF)**: subjects not achieving SVR12 for virologic reasons, including ontreatment failure, ie, viral breakthrough (VBT) or confirmed HCV RNA ≥LLOQ at end of treatment (EOT) for subjects who completed treatment, and viral relapse.

**Non-VF excluded population:** FAS population excluding the subjects who did not achieve SVR12 due to reasons other than VF, including subjects with missing data at the SVR12 time point and subjects who discontinued all treatment prematurely (eg AE or withdrawal of consent).

## 5.3. Virology Time Points and Samples

**Baseline**: the sample taken at baseline or, if not available, the sample taken at screening is used.

**Time of (virologic) failure**: the sample taken at virologic failure (ie at VBT, at actual EOT for subjects with confirmed HCV RNA  $\geq$ LLOQ at EOT or at relapse) with sequencing data available or, if not available, the first available sample after virologic failure with sequencing data available is used.

End of Study (EOS): the last available sample with sequencing data available in the study is used.

### 5.4. Virology Analyses

## 5.4.1. HCV geno/subtype analyses

The number of subjects by HCV geno/subtype for study analyses will be tabulated in frequency outputs (n, %). In addition, a cross-tabulation will compare the HCV geno/subtypes determined at screening (LiPA with NS5B-based reflex) versus baseline (NS5B-based test).

## 5.4.2. Resistance analyses

#### 5.4.2.1. Baseline

The prevalence of baseline polymorphisms, ie the number of subjects with baseline polymorphism, will be tabulated in frequency outputs (n, %) and the amino acid changes from reference at baseline will be listed for all subjects using a 1% cut-off. In addition, subgroup analyses by the presence of baseline polymorphisms may be tabulated to evaluate the impact on response as needed.

#### 5.4.2.2. Post-Baseline

#### Time of Failure

For subjects with failure, the incidence of treatment-emergent and treatment-enriched substitutions will be tabulated (if  $N \ge 10$ ) in frequency outputs (n, %) and the amino acid changes from reference will be listed for all subjects with postbaseline sequencing data using a 1% cut-off.

### **End of Study**

The return to baseline at end of study for the subjects with failure and treatment-emergent substitutions at time of failure will be tabulated (if  $N\ge10$ ) in frequency outputs (n, %) as well as the treatment-emergent substitutions at end of study in the subjects who did not return to baseline.

## 5.4.2.3. Over the Study Period

For the subjects with failure HCV RNA profiles and listings include the reason of failure, relevant baseline disease and demographic characteristics, all amino acid changes from reference at baseline, time of failure and end of study using a 1% cut-off as well as the sequencing follow-up time will be generated. Similar HCV RNA profiles and listings will be generated for subjects with a late viral relapse.

Kaplan-Meier graphs and descriptive statistics will be calculated (if  $N\geq 5$ ) to evaluate the time to return to baseline sequence in subjects with failure and treatment-emergent substitutions at time of failure.

#### 6. SAFETY

Unless specified, all safety analysis will use safety analysis set.

### 6.1. Adverse Events

All reported adverse events (AEs) that are onset during the treatment or follow up phases will be included in the analysis. The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

#### 6.1.1. Definitions

AEs are allocated to the study phases. The phase allocation of AEs consists of a combination of two steps:

- AEs are allocated to phases
- Overlapping/consecutive AEs are combined.

This is detailed in Appendix 1.

**Treatment-emergent Adverse Events (TEAEs)** are AEs that start on or after the first dose or that are a consequence of a preexisting condition that has worsened since baseline.

**AE Duration** is calculated as: AE End date – AE Start date + 1.

**Prevalence**: is defined as the total number of events that occurred (not necessarily new occurrence) in a given time period. The denominator for calculating prevalence and comparable incidence (new occurrences during the same time period) rates will be based on the number of subjects still on treatment at the start of the time period. Note that prevalence counts any AEs regardless whether they are new or sustained from onset prior to the start of the current time interval while comparable incidence refers to new AEs only reported in the current time interval.

## **Events of Special Interest**:

- Cardiac Events
- Increased Bilirubin

#### **Events of Clinical Interest**:

- Rash (all type)
- Photosensitivity conditions
- Pruritus

Note: the search terms for events of special/clinical interest related to MedDRA and MedDRA SMQ are listed in Appendix 2.

## 6.1.2. Analysis Methods

#### **For Adverse Events:**

An overall summary will be provided for all adverse events by treatment cohort for each treatment phase separately (Screening phase, treatment phase, follow-up phase and treatment and follow-up phases). Any AEs, serious AEs, AEs with fatal outcome, AEs by WHO toxicity, treatment related AEs, AEs leading to permanent stop of study medication and relation to HCV infection.

The incidence and the incidence rate of treatment-emergent AEs by system organ class (SOC) and preferred term (PT) will be tabulated for each treatment phase separately (Screening phase, treatment phase, follow-up phase and treatment and follow-up phases). TEAEs in at least 10% of subjects will be tabulated separately,

The incidence and incidence rate of AEs with WHO toxicity grade 3 or 4, SAEs, at least possibly treatment related (AL-335, ODV, and SMV) AEs, AE with fatal outcome and AEs leading to permanent stop of study medication will be tabulated by system organ class (SOC) and preferred term (PT).

The incidence and comparable prevalence rate per 2-week time interval for any AEs will be tabulated to evaluate the safety profile over time (treatment and follow-up phase).

Treatment-emergent AEs will be tabulated by SOC and PT for subgroups: Age and BMI (refer to Section 2.4)

A table will be provided for subjects who met study stopping rules, such as 2nd degree Mobitz Type 2 or 3rd degree heart block, cardiac event that is serious, severe or life-threatening. Drop in LVEF for Echocardiographic(ECHO) by  $\geq$ 10 points with absolute LVEF <50% will be presented too.

Listings will be provided for: all AEs, serious AEs, fatal AEs, AEs leading to permanent stop of AL-335, AEs leading to permanent stop of ODV, AEs leading to permanent stop of SMV andgrade 3-4 AEs. Also AE listing will be provided for the events which meet study stopping rules. AEs which occur in screening will also be included in the listings.

#### For events of interest:

A summary table will be provided for subject incidence with events of interest in treatment and follow-up phases.

The incidence rates of the events of interest by WHO toxicity grades, treatment relationship, with fatal outcome, as an SAE, leading to permanent stop of study medications will be generated in a summary table using frequency and percentage.

The incidence rates will be summarized by PT for each event of interest, and it will be summarized for AEs with worst toxicity grade of 3 or 4 separately as well.

The incidence and prevalence per 2-week time interval will be summarized.

Subgroup analysis by Age, BMI and Gender (refer to Section 2.4) will be conducted for each event of interest by PT.

## 6.2. Clinical Laboratory Tests

Clinical lab data are collected at the screening, baseline, week 1, week 2, week 4, week 6 (BNP only), week 8 (cohort 1), week 10 (cohort 2), EOT, follow up week 4, follow up week 8, follow up week 12, follow up week 18, and follow up week 24 time points.

<u>Baseline</u>: Defined as Day 1 measurement, if available. If not available, then the last assessment before the first administration of study drug will be used.

#### 6.2.1. Definitions

### World Health Organization (WHO) Toxicity grades:

Grades assigned by the central lab will be used. In case no toxicity grades are defined for a test, the abnormalities (above/below normal range) will be used. The abnormalities 'abnormally low' and 'abnormally high' are considered equally important, ie, if a subject has as well an abnormally low as an abnormally high value post baseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%). If, for a specific test, the grading list provides distinct limits for abnormally low (=hypo) values as well as for abnormally high (=hyper) values, this test should be repeated for hyper and hypo limits separately in cross-tabulations and in the ADaM database.

For toxicity grades, no distinction will be made between test results of samples obtained under fasting and under nonfasting conditions: in case limits under fasting and nonfasting conditions differ, the limits of the conditions (fasting/nonfasting) of scheduled visits as planned in the clinical trial protocol (CTP) will always be used, also for samples obtained under a different condition (eg, samples of withdrawal visits).

## **Treatment-emergent:**

An abnormality (toxicity grade or abnormality based on normal ranges) will be considered treatment-emergent if it is worse than the baseline. If the baseline is missing, the abnormality is always considered as treatment-emergent. A shift from 'abnormally low' at baseline to 'abnormally high' post baseline (or vice versa) is also treatment-emergent.

### 6.2.2. Analysis Methods

All analyses will be performed on the treatment and follow-up phases.

Descriptive statistics for the actual values and changes from baseline per timepoint will be performed for all lab parameters with continues values over time by treatment cohort.

Lab toxicity grade and abnormality will be described by frequency and percentage of subjects using below methods:

- Tabulation of the worst treatment-emergent toxicity grade of laboratory parameters
- Tabulation by worst grade of laboratory parameters where at least one subject had worst treatment emergent WHO toxicity grade >=3 during the Treatment Phase
- Cross-tabulation of the worst toxicity grades versus baseline
- Cross-tabulation of toxicity grades versus baseline over time
- Cross-tabulation of the worst laboratory parameter abnormalities versus baseline

Listing is provided for subjects with toxicity grade 3 or greater. The lab results for subjects who had cardiac events will be listed as well.

All analyses will be done on standardized international (SI)-converted values.

## 6.3. Vital Signs and Physical Examination Findings

Vital signs are assessed at following time points: Screening, Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 8, 10 and 12 (10 & 12 for cohort 2), EOT, FU Week 4, and Week 24.

<u>Baseline</u>: Defined as Day 1 measurement, if available. If not available, then the last assessment before the first administration of study drug will be used.

Assessed vital sign parameters are pulse rate, systolic blood pressure (SBP) and diastolic blood pressure (DBP). All measurements should be taken supine and preceded by at least 5 minutes of rest.

#### 6.3.1. Definitions

Pulse rate, SBP and DBP are classified in the following abnormality codes:

**Table 5:** Abnormality Codes for Vital Signs

| | Pulse (bpm) | DBP (mm Hg) | SBP (mm Hg) |
|---------------------|-------------|--------------------|---------------|
| Abnormally low | ≤ 50 | ≤ 50 | ≤ 90 |
| Grade 1 or mild | - | > 90 - < 100 | > 140 - < 160 |
| Grade 2 or moderate | - | $\geq 100 - < 110$ | ≥ 160 - < 180 |
| Grade 3 or severe | - | ≥ 110 | ≥ 180 |
| Abnormally high | ≥ 120 | - | - |

In determining the abnormalities, the following rules are applied:

- The worst grades/abnormalities are determined over the whole observational period (over both the treatment and follow-up phases), including postbaseline scheduled and unscheduled measurements
- The abnormalities 'abnormally low' and 'abnormally high'/grades are considered equally important, ie, if a subject has as well an abnormally low as an abnormally high or graded value postbaseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can be more than 100%)

### **Treatment-emergent:**

An abnormality will be considered treatment-emergent if it is worse than the baseline. If the baseline is missing, the abnormality is always considered as treatment-emergent. A shift from 'abnormally low' at baseline to 'abnormally high' or 'grade ...' post baseline (or vice versa) is also treatment-emergent.

### 6.3.2. Analysis Methods

All analyses will be performed on the treatment and follow-up phases. Vital signs data will be analyzed using descriptive statistics on actual values and change from baseline over time by treatment cohort.

Abnormality of vital signs will be described by frequency and percentage using below methods:

• Tabulation of the worst treatment-emergent abnormality of vital signs

- Tabulation of normality/abnormality of vital signs over time
- Cross-tabulations for the worst abnormality versus baseline

Physical examination data will only be listed.

## 6.4. Electrocardiogram

The electrocardiogram (ECG) variables that will be analyzed are heart rate, PR interval, QRS interval, RR interval, QT interval, and QT interval corrected for heart rate according to Bazett's QT correction (QTcB) and Fridericia's QT correction (QTcF).

ECG data will be collected for the following time points: screening, baseline, day 2, day 3, weeks 1-4, 6, 8, 10 (cohort 2), EOT and follow up week 4. Baseline is the day 1 measurement, if available. If not available, the last assessment before the first administration of study drug will be used.

### 6.4.1. Definitions

For absolute HR, PR and QRS, the following abnormality categories are defined (Table 6).

**Table 6:** Abnormality Categories for ECG

| | HR | PR | QRS |
|-----------------|-----------|----------|----------|
| abnormally low | ≤ 50 bpm | < 120 ms | NAP |
| abnormally high | ≥ 120 bpm | > 200 ms | ≥ 120 ms |

Toxicity grading for PR interval will be performed according to the Division of Aids (DAIDS) grading table for the severity of adult and pediatric adverse events version 1.0, December 2004; clarification August 2009. Please see the Table 7.

**Table 7:** Toxicity Grading for PR Interval

| Parameter | Grade 1<br>Mild | Grade 2<br>Moderate | Grade 3<br>Severe | Grade 4 Potentially life- |
|---|---|---|---|---|
| D 1 1DD 1 | 1 | | | threatening |
| Prolonged PR interva | ıl | | | |
| Adult >16 years | PR interval | PR interval | Type II 2 <sup>nd</sup> degree | Complete AV |
| | 0.20 - 0.25 sec* | >0.25 sec | AV block OR | block |
| | | | Ventricular pause | |
| | | | >3.0 sec | |

<sup>\*</sup>Revised by the sponsor.

The toxicity of PR interval will also be coded using the DAIDS grading table (version 2.0, dated 2014) as follows (http://rsc.tech-res.com/docs/default-source/safety/daids ae grading table v2 nov2014.pdf?sfvrsn=8):

- Grade 1: 210 to <250 msec</li>
- Grade 2: ≥250 msec OR Type I 2nd degree AV block
- Grade 3: Type II 2nd degree AV block OR Ventricular pause ≥3000 msec
- Grade 4: Complete AV block

Analysis for PR will be conducted for all of definitions above (Abnormally high vs low, and toxicity grade per protocol and DAIDS 2.0).

Please note the information for ventricular pause will be provided from medical team.

For absolute QTc parameters the following abnormality categories are defined (based on the ICH E14 Guidance):

- QTc  $\leq$ 450 msec (normal)
- 450 msec <QTc <480 msec (borderline)
- $480 \text{ msec} < \text{QTc} \le 500 \text{ msec (prolonged)}$
- QTc >500 msec (pathologically prolonged).

For increases from baseline in QTc (msec) the following categories are defined (based on ICH E14 Guidance):

- < 30 msec (normal)
- $\geq 30 60$  msec (borderline)
- > 60 msec (abnormally high)

Only increases in QTc  $\geq$ 30 msec will be considered as abnormalities.

In determining the abnormalities, the following rules are applied:

- The worst abnormalities are determined over the whole observational period (over both the treatment and Follow up phases), including postbaseline scheduled and unscheduled measurements.
- The abnormalities 'abnormally low' and 'abnormally high' are considered equally important, ie, if a subject has as well an abnormally low as an abnormally high value postbaseline, both abnormalities are shown in the tables. (This means that the sum of the percentages can by more than 100%)

### **Treatment-emergent:**

An abnormality will be considered treatment-emergent if it is worse than the baseline. If the baseline is missing, the abnormality is always considered as treatment-emergent.

## 6.4.2. Analysis Methods

All analyses will be performed on the treatment and follow-up phases by treatment cohort.

The average of triplicate measurements at each time point will be used for analysis.

Descriptive statistics for the ECG parameters will be calculated for observed values and changes from baseline (CFB) at each scheduled time point.

For individual ECG parameters, the abnormality will be tabulated using frequency and percentage through below methods:

- Tabulation of the worst treatment-emergent ECG abnormalities
- Tabulation of ECG normality/abnormalities over time
- Cross-Tabulation of the Worst ECG Abnormalities in Actual Value versus baseline value
- Cross-Tabulation of the Worst QTc Increase versus the abnormality on the actual value

A listing of ECG abnormalities (all parameters) will be provided. It will contain both actual and CFB values.

## 6.5. Echocardiography

Echocardiographic (ECHO) data will include Left Ventricular (LV) Ejection Fraction (LVEF) in percent (%). Additional parameters include:

- Systolic Volume (mL)
- Diastolic Volume (mL)
- LV Fractional Shortening (%)
- LV Posterior Wall (PW) Diastolic Thickness (cm)
- Ventricular Septum Diastolic Thickness (cm)

ECHO data will be collected in the following time points: screening, week 4, week 8, EOT, follow up week 4. The last assessment before the first administration of study drug will be used as the baseline.

#### 6.5.1. Definitions

The following definitions are applicable to the ECHO analyses:

- Reversible decrease in LVEF is defined as a decrease of >10% from baseline, which is followed by an increase or a decrease of <=5% from baseline.
- No resolution in LVEF is defined as a decrease of >10% from baseline, which is not followed by an increase or a decrease of <=5% from baseline.

## 6.5.2. Analysis Methods

All analyses will be performed over the treatment and follow-up phases by treatment cohort.

Descriptive statistics for the ECHO parameters will be calculated for observed values and changes from baseline at each scheduled time point. Number and percent of subjects abnormally low, normal, and abnormally high ECHO parameters by week of study will be summarized for each ECHO parameter.

Number and percentage of subjects with a maximum LVEF change from baseline over all postbaseline visits will be reported for the following categories: decline of >10%, decline of >5 -

 $\leq$ 10%, decline of  $\leq$ =5%, increase of >5 - <=10%, increase of >10%, and increase of <5%. Each of the following will also be summarized: The number and percentage of subjects with a maximum decline of baseline over all postbaseline visits of >10% AND:

- Resulting in a LVEF% of <50%.
- A maximum decline of baseline of >10% with reversible decrease.
- A maximum decline of baseline of >10% with no resolution.

And the time to onset for LVEF decrease and duration will also be summarized.

Number and percentage of subjects will be summarized by postbaseline visit for subjects who have a decrease in LVEF of:

- >5% but  $\leq 10\%$
- >10%

A listing of ECHO with actual value, change from baseline, or all parameters will be provided.

#### 6.6. Patient Profiles

A set of patient profiles will be produced for each subject. Data presented will include baseline characteristics, medical history, disposition, study drug exposure, adverse events, HCV RNA levels, lab parameters, ECG parameters, and concomitant medications. Lab parameters will include Bilirubin (all version), AST, ALT, ALP, GGT, Creatine Kinase, Amylase, Lipase, BNP, e-GFR.

### 7. PHARMACOKINETICS/PHARMACODYNAMICS

Pharmacokinetic (PK) analysis and Pharmacokinetic/Pharmacodynamic analysis will be performed by PK analysis vender and results will be reported by PK analysis vender. Pharmacodynamic (PD) analysis is not planned.

#### 7.1. Pharmacokinetics

Details of the analysis plan and summary of results from Pharmacokinetic analyses will be provided in a separate report by PK analysis vender.

### 7.2. Immune Response

Not applicable.

## 7.3. Pharmacodynamics

PD analysis is not planned.

## 7.4. Pharmacokinetic/Pharmacodynamic Relationships

The Pharmacokinetic/Pharmacodynamic relationship of plasma concentrations and ECG parameters will be evaluated. Details of the analysis plan and summary of results from Pharmacokinetic/Pharmacodynamic analyses will be provided in a separate report.

### **ATTACHMENTS**

#### **APPENDIX 1: PHASE ALLOCATION/COMBINING AES**

## STEP 1: allocation of events to the phases

Adverse events present in the SDS database are allocated to phases based on their start date. If the start date of an event falls between (or on) the start and stop date of a phase, the AE is attributed to that phase.

Incomplete dates (ie, day and/or month and/or year missing)

## • Partial start or stop dates:

- 1. The partial start date (ie, missing day) will be imputed with the first day of the month unless the month/year is the same as the month/year of an analysis phase. In this situation the incomplete start date will be imputed with the start date of that phase. If the start date of the year is given without specification of the month and date, the partial missing start date will be imputed with the maximum of the first day of the given year and the first date of the first phase.
- 2. The partial missing end date (ie, missing day) will be imputed with the last day of the month. If the end date of the year is given without specification of the month and date, the partial missing end date will be imputed with the minimum of the last day of the given year and the end date of the last phase.
- <u>Completely missing start date:</u> the event is allocated to the first active treatment phase (the start date is imputed with the treatment phase start date), except if the end date of the AE falls before the start of the first active treatment phase, in which case it is assigned to the screening phase (the start date is imputed with the screening phase start date).
- Completely missing end date: the following decision rules apply
  - 1. For completed and discontinued subjects:
    - In case the end date is not flagged as ongoing the date will remain missing.
    - In case the end date is flagged as ongoing the date is imputed by the end date of the last phase.
  - 2. For ongoing subjects:
    - Missing end dates are imputed by the end date of the last phase (ie, the cut-off date).

#### **STEP 2: combining adverse events**

Overlapping/consecutive events are defined as events of the same subject with the same preferred term who have at least 1 day in overlap or for which the start date of an event is 1 day after the end date of the preceding event. Overlapping/consecutive events may be combined into one AE or not, according to the following rules:

- 1. In case a nonactive phase (eg, Screening) is followed by an active phase, and the overlapping/consecutive events start in both phases, they are allocated to their respective phase and are considered as separate events.
- 2. In case overlapping/consecutive events start within a single phase, they are considered as one and the same AE. The individual events who contribute to this AE are retained as individual records in the ADAM database but are assigned the same onset, phase, and total duration.
- 3. In case an active phase is followed by a nonactive phase (eg, Follow-Up), and the overlapping/consecutive events start in both phases, they are allocated to the active phase and are considered as one and the same AE. The individual events who contribute to this AE are retained as individual records in the ADAM database but are assigned the same duration, onset and active phase.
- 4. In case a nonactive phase is followed by a nonactive phase, and the overlapping/consecutive events start in both phases, they are allocated to their respective phase and are considered as separate AEs.

Events can only be combined into one and the same AE if their start and stop dates are complete. In case the completely missing end date is imputed, this date is also considered as a complete date.

31

## APPENDIX 2A: SEARCH TERMS FOR EVENTS OF SPECIAL/CLINICAL INTEREST

| | MedrDRA Term | Searching Terms |
|---|---|---|
| Events of special interest | Level | |
| Cardiac Events | SMQ | Please see Appendix 3 |
| Increased Bilirubin | MedDRA PTs | Bilirubin conjugated abnormal |
| mereuseu Biniusin | Wied Brain 19 | Bilirubin conjugated increased |
| | | Bilirubin excretion disorder |
| | | Bilirubinuria |
| | | Blood bilirubin abnormal |
| | | Blood bilirubin increased |
| | | Blood bilirubin unconjugated increased |
| | | Hyperbilirubinaemia |
| | | Icterus index increased |
| | | Jaundice |
| | | Jaundice cholestatic |
| | | Jaundice extrahepatic obstructive |
| | | Jaundice hepatocellular |
| | | Ocular icterus |
| | | Urine bilirubin increased |
| | | Yellow skin |
| Events of clinical interest | | |
| Rash (all type) | MedDRA HLTs, | Erythemas - HLT |
| | PTs | Papulosquamous conditions - HLT |
| | | Rashes, eruptions and exanthems NEC - HLT |
| | | PT: |
| | | Photodermatosis |
| | | Photosensitivity reaction |
| | | Polymorphic light eruption |
| | | Solar dermatitis |
| | | Sunburn |
| | SMQ | SMQ-Severe cutaneous adverse reaction: narrow |
| | | scope and selected terms of the broad scope(refer |
| | | Appendix 3) |
| Pruritus | MedDRA HLT | Pruritus NEC |
| | | Photodermatosis |
| | 16 100 : 55 | Photosensitivity reaction |
| Photosensitivity conditions | MedDRA PTs | Polymorphic light eruption |
| | | Solar dermatitis |
| | | Sunburn |

## APPENDIX 2B: RASH - SMQ19.1

SMQ 19.1: "Severe cutaneous adverse reaction"

| SCOPE | Preferred Term |
|--------|----------------------------------------------|
| NARROW | CUTANEOUS VASCULITIS |
| NARROW | DERMATITIS BULLOUS |
| NARROW | DERMATITIS EXFOLIATIVE |
| NARROW | DERMATITIS EXFOLIATIVE GENERALISED |
| NARROW | ERYTHEMA MULTIFORME |
| NARROW | OCULOMUCOCUTANEOUS SYNDROME |
| NARROW | SKIN NECROSIS |
| NARROW | STEVENS-JOHNSON SYNDROME |
| NARROW | TOXIC EPIDERMAL NECROLYSIS |
| NARROW | ACUTE GENERALISED EXANTHEMATOUS PUSTULOSIS |
| NARROW | TOXIC SKIN ERUPTION |
| NARROW | EPIDERMAL NECROSIS |
| NARROW | EXFOLIATIVE RASH |
| NARROW | DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC |
| | SYMPTOMS |
| BROAD | BLISTER |
| BROAD | BULLOUS IMPETIGO |
| BROAD | DRUG ERUPTION |
| BROAD | EPIDERMOLYSIS BULLOSA |
| BROAD | MUCOCUTANEOUS ULCERATION |
| BROAD | NIKOLSKY'S SIGN |
| BROAD | PEMPHIGOID |
| BROAD | PEMPHIGUS |
| BROAD | SKIN EROSION |
| BROAD | SKIN EXFOLIATION |
| BROAD | EPIDERMOLYSIS |
| BROAD | ACQUIRED EPIDERMOLYSIS BULLOSA |

33

## **APPENDIX 3: CARDIAC EVENTS - SMQ19.1**

| | Narrow/Broad | PT Term |
|---|---|---|
| diac arrhythn | | |
| Arrhythmia r | | s, signs and symptoms (SMQ) |
| | Narrow | Chronotropic incompetence |
| | Narrow | Electrocardiogram repolarisation abnormality |
| | Narrow | Electrocardiogram RR interval prolonged |
| | Narrow | Electrocardiogram U-wave abnormality |
| | Narrow | Sudden cardiac death |
| | Broad | Bezold-Jarisch reflex |
| | Broad | Bradycardia |
| | Broad | Cardiac arrest |
| | Broad | Cardiac death |
| | Broad | Cardiac telemetry abnormal |
| | Broad | Cardio-respiratory arrest |
| | Broad | Central bradycardia |
| | Broad | Electrocardiogram abnormal |
| | Broad | Electrocardiogram ambulatory abnormal |
| <del> </del> | Broad | Electrocardiogram change |
| ++++ | Broad | Heart rate abnormal |
| +++ | Broad | Heart rate decreased |
| <del>- </del> | Broad | Heart rate increased |
| + + + | Broad | Loss of consciousness |
| | Broad | Palpitations |
| | Broad | Rebound tachycardia |
| | Broad | Sudden death |
| | Broad | Syncope |
| +++ | Broad | |
| | | Tachycardia paroxyamal |
| | Broad | Tachycardia paroxysmal |
| Cardiac arrhy | Broad<br>ythmia terms (incl b | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) |
| Cardiac arrhy<br>Bradyarr | Broad<br>ythmia terms (incl b | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) |
| Cardiac arrhy<br>Bradyarr<br>(SMQ) | Broad<br>ythmia terms (incl b<br>hythmias (incl cond | Tachycardia paroxysmal<br>oradyarrhythmias and tachyarrhythmias) (SMQ)<br>uction defects and disorders of sinus node function |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad<br>ythmia terms (incl b<br>hythmias (incl cond<br>lyarrhythmia terms | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function, nonspecific (SMQ) |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad<br>ythmia terms (incl b<br>hythmias (incl cond<br>lyarrhythmia terms<br>Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function , nonspecific (SMQ) Bradyarrhythmia |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function , nonspecific (SMQ) Bradyarrhythmia Ventricular asystole |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function , nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function, nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow Narrow Narrow Narrow Narrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow Narrow Narrow Narrow Narrow Narrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation |
| Cardiac arrhy Bradyarr (SMQ) Brad | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal pradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node functions, nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function , nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function , nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow Marrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node functions. nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block Brugada syndrome |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block Brugada syndrome |
| Cardiac arrhy Bradyarr (SMQ) Brad Cond | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow duction defects (SM Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block Brugada syndrome Bundle branch block |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow Marrow Narrow | Tachycardia paroxysmal oradyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block Brugada syndrome Bundle branch block Bundle branch block bilateral |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow Marrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Bifascicular block Brugada syndrome Bundle branch block Bundle branch block left |
| Cardiac arrhy Bradyarr (SMQ) Brad Cone | Broad ythmia terms (incl b hythmias (incl cond lyarrhythmia terms Narrow Narrow Marrow Narrow | Tachycardia paroxysmal radyarrhythmias and tachyarrhythmias) (SMQ) uction defects and disorders of sinus node function nonspecific (SMQ) Bradyarrhythmia Ventricular asystole Q) Accessory cardiac pathway Adams-Stokes syndrome Agonal rhythm Atrial conduction time prolongation Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular dissociation Bifascicular block Brugada syndrome Bundle branch block Bundle branch block left Bundle branch block right |

| | Nomery/Dreed | DT Torres |
|---|---|---|
| | Narrow/Broad Narrow | PT Term Electrocardio grow PO interval prolonged |
| | | Electrocardiogram PQ interval prolonged |
| | Narrow | Electrocardiogram PQ interval shortened |
| | Narrow | Electrocardiogram PR prolongation |
| | Narrow | Electrocardiogram PR shortened |
| | Narrow | Electrocardiogram QRS complex prolonged |
| | Narrow | Electrocardiogram QT prolonged |
| | Narrow | Electrocardiogram repolarisation abnormality |
| | Narrow | Lenegre's disease |
| | Narrow | Long QT syndrome |
| | Narrow | Paroxysmal atrioventricular block |
| _ | Narrow | Sinoatrial block |
| | Narrow | Trifascicular block |
| | Narrow | Ventricular dyssynchrony |
| | Narrow | Wolff-Parkinson-White syndrome |
| | Disorders of sinus no | |
| | Narrow | Nodal arrhythmia |
| | Narrow | Nodal rhythm |
| | Narrow | Sinus arrest |
| | Narrow | Sinus arrhythmia |
| | Narrow | Sinus bradycardia |
| | Narrow | Sinus node dysfunction |
| | Narrow | Wandering pacemaker |
| | Cardiac arrhythmia terms | |
| | Narrow | Arrhythmia |
| | Narrow | Heart alternation |
| | Narrow | Heart rate irregular |
| | Narrow | Pacemaker generated arrhythmia |
| | Narrow | Pacemaker syndrome |
| | Narrow | Paroxysmal arrhythmia |
| | Narrow | Pulseless electrical activity |
| | Narrow | Reperfusion arrhythmia |
| | Narrow | Withdrawal arrhythmia |
| | | praventricular and ventricular tachyarrhythmias) |
| | (SMQ) | |
| | | hyarrhythmias (SMQ) |
| | | Arrhythmia supraventricular |
| | Narrow | Atrial fibrillation |
| | Narrow | Atrial flutter |
| $\perp$ | Narrow | Atrial parasystole |
| | Narrow | Atrial tachycardia |
| | Narrow | Junctional ectopic tachycardia |
| $\perp$ | Narrow | Sinus tachycardia |
| $\perp$ | Narrow | Supraventricular extrasystoles |
| | Narrow | Supraventricular tachyarrhythmia |
| $\perp$ | Narrow | Supraventricular tachycardia |
| | Broad | ECG P wave inverted |
| | Broad | Electrocardiogram P wave abnormal |
| | Broad | Retrograde p-waves |
| _ | The state of the s | ms, nonspecific (SMQ) |
| $\perp$ | Narrow | Anomalous atrioventricular excitation |
| | Narrow | Cardiac fibrillation |
| | Narrow | Cardiac flutter |
| | Narrow | Extrasystoles |
| | Narrow | Tachyarrhythmia |

| | NI /D 1 | DOT OF |
|---|---|---|
| | Narrow/Broad | PT Term |
| Ve | ntricular tachyarrhy | |
| | Narrow | Accelerated idioventricular rhythm |
| | Narrow | Cardiac fibrillation |
| | Narrow | Parasystole |
| | Narrow | Rhythm idioventricular |
| | Narrow | Torsade de pointes |
| | Narrow | Ventricular arrhythmia |
| | Narrow | Ventricular extrasystoles |
| | Narrow | Ventricular fibrillation |
| | Narrow | Ventricular flutter |
| | Narrow | Ventricular parasystole |
| | Narrow | Ventricular pre-excitation |
| | Narrow | Ventricular tachyarrhythmia |
| | Narrow | Ventricular tachycardia |
| Cardiac failure | <del>-</del> / | |
| | Narrow | Acute left ventricular failure |
| | Narrow | Acute pulmonary oedema |
| | Narrow | Acute right ventricular failure |
| | Narrow | Cardiac asthma |
| | Narrow | Cardiac failure |
| | Narrow | Cardiac failure acute |
| | Narrow | Cardiac failure chronic |
| | Narrow | Cardiac failure congestive |
| | Narrow | Cardiac failure high output |
| | Narrow | Cardiogenic shock |
| | Narrow | Cardiopulmonary failure |
| | Narrow | Cardiorenal syndrome |
| | Narrow | Chronic left ventricular failure |
| | Narrow | Chronic right ventricular failure |
| | Narrow | Cor pulmonale |
| | Narrow | Cor pulmonale acute |
| | Narrow | Cor pulmonale chronic |
| | Narrow | Ejection fraction decreased |
| | Narrow | Hepatic congestion |
| | Narrow | Hepatojugular reflux |
| | Narrow | Left ventricular failure |
| | Narrow | Low cardiac output syndrome |
| | Narrow | Neonatal cardiac failure |
| | Narrow | Obstructive shock |
| | Narrow | Pulmonary oedema |
| | Narrow | Pulmonary oedema neonatal |
| | Narrow | Radiation associated cardiac failure |
| | Narrow | Right ventricular ejection fraction decreased |
| | Narrow | Right ventricular failure |
| | Narrow | Ventricular failure |
| | Broad | Artificial heart implant |
| | Broad | Atrial natriuretic peptide abnormal |
| | Broad | Atrial natriuretic peptide increased |
| | Broad | Bendopnoea |
| | Broad | Brain natriuretic peptide abnormal |
| | Broad | Brain natriuretic peptide increased |
| | Broad | Cardiac cirrhosis |
| | Broad | Cardiac contractility modulation therapy |
| | Broad | Cardiac index decreased |

| | D. J. DELT |
|---|---|
| Narrow/ | |
| Broad | Cardiac output decreased |
| Broad | Cardiac resynchronisation therapy |
| Broad | Cardiac ventriculogram abnormal |
| Broad | Cardiac ventriculogram left abnormal |
| Broad | Cardiac ventriculogram right abnormal |
| Broad | Cardiomegaly |
| Broad | Cardio-respiratory distress Cardiothoracic ratio increased |
| Broad | |
| Broad | Central venous pressure increased |
| Broad | Diastolic dysfunction Dilatation ventricular |
| Broad | |
| Broad | Dyspnoea paroxysmal nocturnal |
| Broad | Heart transplant |
| Broad | Hepatic vein dilatation |
| Broad | Jugular vein distension |
| Broad | Left ventricular dilatation |
| Broad | Left ventricular dysfunction |
| Broad | Left ventricular enlargement |
| Broad | Lower respiratory tract congestion |
| Broad | Myocardial depression |
| Broad | Nocturnal dyspnoea |
| Broad | N-terminal prohormone brain natriuretic peptide |
| | abnormal |
| Broad | N-terminal prohormone brain natriuretic peptide |
| | increased |
| Broad | Oedema |
| Broad | Oedema due to cardiac disease |
| Broad | Oedema neonatal |
| Broad | Oedema peripheral |
| Broad | Orthopnoea |
| Broad | Peripheral oedema neonatal |
| Broad | Peripheral swelling |
| Broad | Post cardiac arrest syndrome |
| Broad | Prohormone brain natriuretic peptide abnormal |
| Broad | Prohormone brain natriuretic peptide increased |
| Broad | Pulmonary congestion |
| Broad | Right ventricular dilatation |
| Broad | Right ventricular dysfunction |
| Broad | Right ventricular enlargement |
| Broad | Scan myocardial perfusion abnormal |
| Broad | Stroke volume decreased |
| Broad | Surgical ventricular restoration |
| Broad | Systolic dysfunction |
| Broad | Venous pressure increased |
| Broad | Venous pressure jugular abnormal |
| Broad | Venous pressure jugular increased |
| Broad | Ventricular assist device insertion |
| Broad | Ventricular dysfunction |
| Broad | Ventricular dyssynchrony |
| Cardiomyopathy (SMQ) | |
| Narrow | Atrial septal defect acquired |
| Narrow | Biopsy heart abnormal |
| Narrow | Cardiac amyloidosis |
| Narrow | Cardiac hypertrophy |

| Narrow/Broad | PT Term |
|---|---|
| Narrow | Cardiac sarcoidosis |
| Narrow | Cardiac septal hypertrophy |
| Narrow | Cardiac siderosis |
| Narrow | Cardiomyopathy |
| Narrow | Cardiomyopathy acute |
| Narrow | Cardiomyopathy alcoholic |
| Narrow | Cardiomyopathy neonatal |
| Narrow | Cardiotoxicity |
| Narrow | Congestive cardiomyopathy |
| Narrow | Cytotoxic cardiomyopathy |
| Narrow | Diabetic cardiomyopathy |
| Narrow | Ejection fraction abnormal |
| Narrow | Ejection fraction decreased |
| Narrow | Eosinophilic myocarditis |
| Narrow | HIV cardiomyopathy |
| Narrow | Hypertensive cardiomyopathy |
| Narrow | Hypertrophic cardiomyopathy |
| Narrow | Ischaemic cardiomyopathy |
| Narrow | Metabolic cardiomyopathy |
| Narrow | Myocardial calcification |
| Narrow | Myocardial fibrosis |
| Narrow | Myocardial haemorrhage |
| Narrow | Non-obstructive cardiomyopathy |
| Narrow | Peripartum cardiomyopathy |
| Narrow | Pulmonary arterial wedge pressure increased |
| Narrow | Restrictive cardiomyopathy |
| Narrow | Right ventricular ejection fraction decreased |
| Narrow | Stress cardiomyopathy |
| Narrow | Tachycardia induced cardiomyopathy |
| Narrow | Thyrotoxic cardiomyopathy |
| Narrow | Ventricular septal defect acquired |
| Narrow | Viral cardiomyopathy |
| Broad | Abnormal precordial movement |
| Broad | Acquired cardiac septal defect |
| Broad | Acute left ventricular failure |
| Broad | Alcohol septal ablation |
| Broad | Allergic myocarditis |
| Broad | Arrhythmia |
| Broad | Arrhythmia supraventricular |
| Broad | Artificial heart implant |
| Broad | Ascites |
| Broad | Atrial hypertrophy |
| Broad | Atrial pressure increased |
| Broad | Autoimmune myocarditis |
| Broad | Bendopnoea |
| Broad | Blood pressure diastolic abnormal |
| Broad | Blood pressure diastolic decreased |
| Broad | Blood pressure diastolic increased |
| Broad | Blood pressure fluctuation |
| Broad | Blood pressure inadequately controlled |
| Broad<br>Broad | Blood pressure systolic abnormal |
| Broad | Blood pressure systolic decreased Blood pressure systolic increased |
| Broad | Cardiac aneurysm |
| DIVau | Cardiac anedrysin |

| T | |
|--------------|-------------------------------------------|
| Narrow/Broad | PT Term |
| Broad | Cardiac arrest |
| Broad | Cardiac contractility modulation therapy |
| Broad | Cardiac electrophysiologic study abnormal |
| Broad | Cardiac failure |
| Broad | Cardiac failure acute |
| Broad | Cardiac failure chronic |
| Broad | Cardiac failure congestive |
| Broad | Cardiac function test abnormal |
| Broad | Cardiac imaging procedure abnormal |
| Broad | Cardiac index abnormal |
| Broad | Cardiac index decreased |
| Broad | Cardiac index increased |
| Broad | Cardiac monitoring abnormal |
| Broad | Cardiac operation |
| Broad | Cardiac output decreased |
| Broad | Cardiac pseudoaneurysm |
| Broad | Cardiac resynchronisation therapy |
| Broad | Cardiac ventricular scarring |
| Broad | Cardiac ventriculogram abnormal |
| Broad | Cardiac ventriculogram left abnormal |
| Broad | Cardiac ventriculogram right abnormal |
| Broad | Cardiomegaly |
| Broad | Cardiothoracic ratio increased |
| Broad | Cardiovascular disorder |
| Broad | Cardiovascular function test abnormal |
| Broad | Chest pain |
| Broad | Chest X-ray abnormal |
| Broad | Computerised tomogram thorax abnormal |
| Broad | Coxsackie carditis |
| Broad | Coxsackie myocarditis |
| Broad | Cytomegalovirus myocarditis |
| Broad | Decreased ventricular preload |
| Broad | Diastolic dysfunction |
| Broad | Dilatation atrial |
| Broad | Dilatation ventricular |
| Broad | Directional Doppler flow tests abnormal |
| Broad | Dyspnoea |
| Broad | ECG signs of ventricular hypertrophy |
| Broad | Echocardiogram abnormal |
| Broad | Electrocardiogram abnormal |
| Broad | Electrocardiogram change |
| Broad | Endocardial fibroelastosis |
| Broad | External counterpulsation |
| Broad | Gonococcal heart disease |
| Broad | Heart and lung transplant |
| Broad | Heart transplant |
| Broad | Hepatomegaly |
| Broad | Hyperdynamic left ventricle |
| Broad | Increased ventricular preload |
| Broad | Irregular breathing |
| Broad | Labile blood pressure |
| Broad | Left atrial dilatation |
| Broad | Left atrial enlargement |
| Broad | Left ventricular dilatation |

| Narrow/Broad | PT Term |
|---|---|
| Broad | Left ventricular end-diastolic pressure decreased |
| Broad | Left ventricular enlargement |
| Broad | Left ventricular failure |
| Broad | Left ventricular heave |
| Broad | Lupus myocarditis |
| Broad | Lyme carditis |
| Broad | Malarial myocarditis |
| Broad | Mental status changes |
| Broad | Multiple gated acquisition scan abnormal |
| Broad | Myocardiac abscess |
| Broad | Myocardial necrosis marker increased |
| Broad | Myocarditis |
| Broad | Myocarditis bacterial |
| Broad | Myocarditis helminthic |
| Broad | Myocarditis infectious |
| Broad | Myocarditis meningococcal |
| Broad | Myocarditis mycotic |
| Broad | Myocarditis post infection |
| Broad | Myocarditis septic |
| Broad | Myocarditis syphilitic |
| Broad | Myocarditis toxoplasmal |
| Broad | Myoglobinaemia |
| Broad | Myoglobinuria |
| Broad | Nocturia |
| Broad | Nuclear magnetic resonance imaging thoracic |
| | abnormal |
| Broad | Oedema |
| Broad | Orthostatic hypotension |
| Broad | Palpitations |
| Broad | Papillary muscle disorder |
| Broad | Papillary muscle haemorrhage |
| Broad | Radiation myocarditis |
| Broad | Right atrial dilatation |
| Broad | Right atrial enlargement |
| Broad | Right atrial pressure increased |
| Broad | Right ventricle outflow tract obstruction |
| Broad | Right ventricular dilatation |
| Broad<br>Broad | Right ventricular enlargement Right ventricular heave |
| Broad | Right ventricular neave Right ventricular systolic pressure decreased |
| Broad | Scan myocardial perfusion abnormal |
| Broad | Sudden cardiac death |
| Broad | Sudden death Sudden death |
| Broad | Surgical ventricular restoration |
| Broad | Syncope Syncope |
| Broad | Systolic anterior motion of mitral valve |
| Broad | Systolic dysfunction |
| Broad | Ultrasound Doppler abnormal |
| Broad | Vascular resistance pulmonary increased |
| Broad | Ventricular arrhythmia |
| Broad | Ventricular assist device insertion |
| Broad | Ventricular dysfunction |
| Broad | Ventricular dyskinesia |
| Broad | Ventricular dyssynchrony |
| <br>i e | , |

| 1 | Narrow/Broad | PT Term |
|---|---|---|
| | Broad | Ventricular hyperkinesia |
| | Broad | Ventricular hyperkniesia Ventricular hyperkniesia |
| | Broad | Ventricular hypothophy Ventricular hypothophy |
| | Broad | Ventricular remodelling |
| | Broad | Viral myocarditis |
| Ischaemic heart di | | virai myocardius |
| Myocardial inf | | |
| | Varrow | Acute coronary syndrome |
| | Varrow | Acute myocardial infarction |
| | Varrow | Angina unstable |
| | Narrow | Blood creatine phosphokinase MB abnormal |
| | Varrow | Blood creatine phosphokinase MB increased |
| | Varrow | Coronary artery embolism |
| | Narrow | Coronary artery occlusion |
| | Narrow | Coronary artery reocclusion |
| | Narrow | Coronary artery thrombosis |
| | Narrow<br>Narrow | Coronary bypass thrombosis Coronary vascular graft occlusion |
| | Narrow<br>Narrow | Kounis syndrome |
| | | ř |
| | Narrow | Myocardial infarction Myocardial necrosis |
| | Narrow | J |
| | Narrow | Myocardial reperfusion injury |
| | Narrow | Myocardial stunning |
| | Narrow | Papillary muscle infarction |
| | Narrow | Post procedural myocardial infarction |
| | Narrow | Postinfarction angina |
| | Narrow | Silent myocardial infarction |
| | Narrow | Troponin I increased |
| | Narrow | Troponin increased |
| | Narrow | Troponin T increased |
| | Broad | Blood creatine phosphokinase abnormal |
| | Broad | Blood creatine phosphokinase increased |
| | Broad | Cardiac ventricular scarring |
| | Broad | ECG electrically inactive area |
| | Broad | ECG signs of myocardial infarction |
| | Broad | Electrocardiogram Q wave abnormal |
| | Broad | Electrocardiogram ST segment abnormal |
| | Broad | Electrocardiogram ST segment elevation |
| | Broad | Electrocardiogram ST-T segment elevation |
| | Broad | Infarction |
| | Broad | Myocardial necrosis marker increased |
| | Broad | Scan myocardial perfusion abnormal |
| | Broad | Vascular graft occlusion |
| | Broad | Vascular stent occlusion |
| | Broad | Vascular stent thrombosis |
| Shock (SMQ) | | |
| | | ardiac conditions (excl torsade de pointes) (SMQ) |
| | Varrow | Acute left ventricular failure |
| | Varrow | Adams-Stokes syndrome |
| | Varrow | Atrial parasystole |
| | Varrow | Cardiac arrest |
| | Varrow | Cardiac arrest neonatal |
| | Varrow | Cardiac death |
| 1 | Narrow | Cardiac fibrillation |

| | | <b>y</b> |
|---|---|---|
| | Narrow/Broad | PT Term |
| | Narrow | Cardiac flutter |
| | Narrow | Cardiogenic shock |
| | Narrow | Cardio-respiratory arrest |
| | Narrow | Cardio-respiratory arrest neonatal |
| | Narrow | Cardiovascular insufficiency |
| - | Narrow | Circulatory collapse |
| | Narrow | Obstructive shock |
| | Narrow | Pulse absent |
| | Narrow | Pulseless electrical activity |
| | | • |
| | Narrow | Shock |
| | Narrow | Shock symptom |
| | Narrow | Sudden cardiac death |
| | Narrow | Ventricular asystole |
| | Narrow | Ventricular fibrillation |
| | Narrow | Ventricular flutter |
| | Narrow | Ventricular parasystole |
| | Broad | Acute kidney injury |
| | Broad | Acute prerenal failure |
| | Broad | Acute respiratory failure |
| | Broad | Anuria |
| | Broad | Blood pressure immeasurable |
| | Broad | Cerebral hypoperfusion |
| | Broad | Grey syndrome neonatal |
| | Broad | Hepatic congestion |
| | Broad | Hepatojugular reflux |
| | Broad | Hepatorenal failure |
| | Broad | Hypoperfusion |
| | Broad | Jugular vein distension |
| | Broad | Myocardial depression |
| | Broad | Neonatal anuria |
| | Broad | Neonatal multi-organ failure |
| | Broad | Neonatal respiratory failure |
| | Broad | Organ failure |
| | Broad | Prerenal failure |
| | Broad | Propofol infusion syndrome |
| | Broad | Renal failure |
| | Broad | Renal failure neonatal |
| | Broad<br>es/QT prolongation ( | Respiratory failure |
| | Narrow | Electrocardiogram QT interval abnormal |
| | Narrow | Electrocardiogram QT prolonged |
| | Narrow | Long QT syndrome |
| | Narrow | Long QT syndrome congenital |
| | Narrow<br>Narrow | Torsade de pointes Ventricular tachycardia |
| | Broad | Cardiac arrest |
| | Broad | Cardiac death |
| | Broad | Cardiac death Cardiac fibrillation |
| | Broad | Cardio-respiratory arrest |
| | Broad | Electrocardiogram repolarisation abnormality |
| | Broad | |
| | | Electrocardiogram U-wave abnormality Loss of consciousness |
| | Broad | Sudden cardiac death |
| | Broad | |
| | Broad | Sudden death |

# NCT02993250

## AL-335, Odalasvir, TMC435(simeprevir)

## Statistical Analysis Plan 64294178HPC2003

| Narrow/Broad | PT Term | |
|--------------|---------|-----------------------------|
| | Broad | Syncope |
| | Broad | Ventricular arrhythmia |
| | Broad | Ventricular fibrillation |
| | Broad | Ventricular flutter |
| | Broad | Ventricular tachyarrhythmia |